CLINICAL TRIAL: NCT01694615
Title: Prospective Controlled Study of Transbronchial Cryoprobe Versus Forceps Biopsy for Acute Rejection in Lung Transplantation
Brief Title: Cryoprobe Transbronchial Lung Biopsy in Lung Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NA_00052081
Record Dates: First submitted 2012-09-17; First posted 2012-09-27 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Lung Transplantation
Keywords: Lung Transplantation; Acute Rejection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cryoprobe biopsy (Active Comparator): All patients enrolled will undergo standard forceps biopsies followed by cryoprobe biopsies and results will be compared
  Interventions: Procedure: Cryoprobe biopsy
- Forceps Biopsy (Active Comparator): All patients enrolled will undergo standard forceps biopsies followed by cryoprobe biopsies and results will be compared
  Interventions: Procedure: Forceps Biopsy

INTERVENTIONS:
Procedure: Cryoprobe biopsy
  Arms: Cryoprobe biopsy
Procedure: Forceps Biopsy
  Arms: Forceps Biopsy

SUMMARY:
Lung transplant recipients undergo bronchoscopy with biopsies for clinical indications and for surveillance in the diagnosis of acute rejection using standard transbronchial forceps. It is recognized that standard forceps biopsies underestimate the presence or degree of airway rejection due to crush artifact and sample size. Transbronchial cryobiopsies have been shown in the literature to provide larger samples without crush artifact in a safe fashion in lung cancer patients. The aim of this study is to determine if transbronchial cryobiopsy is superior to standard transbronchial forceps biopsies in regards to sample size, architecture and the diagnosis of early rejection in lung transplant recipients which if discovered earlier may improve survival.

ELIGIBILITY:
Inclusion Criteria:

* Individuals referred for either clinically indicated or surveillance flexible bronchoscopy will be included in the study population
* Age greater than 18 years and having undergone bilateral orthotopic lung transplantation

Exclusion Criteria:

* Coagulopathy: plts < 50,000 international normalized ratio (INR) > 1.5
* Forced expiratory volume at one second (FEV1) < 0.8
* Diffuse bullous disease
* Hemodynamic instability
* Severe hypoxemia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Differences in size of biopsy specimen and architectural preservation of the airways/alveoli (ie degree of crush artifact) | From date of study enrollment until the patient is 2 years post lung transplant
  Direct measurements of pathologic specimens from the forceps and cryoprobe will be compared. In addition, amount of crush artifact will alse be directly measured and compared utilizing pathology software which measures area of viable tissue.

SECONDARY OUTCOMES:
Diagnostic yield (ie presence of acute cellular rejections (ACR), chronic rejection, lymphocytic bronchiolitis and infection) | From date of study enrollment until the patient is 2 years post lung transplant
  Each specimen will be independently reviewed by a lung transplant pathology physician to determine the presence or absence of rejection and results compared. All data will be available to the transplant team in the event any rejection is found, it will be acted upon immediately as per the transplant teams protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Lonny Yarmus, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States